CLINICAL TRIAL: NCT05401682
Title: Prospective Study of Post Surgical Continued Pain (PSCP) Patients Undergoing Flexion Distraction Decompression Spinal Manipulation
Brief Title: Prospective Study of Post Surgical Continued Spinal Pain Patients
Status: Completed | Type: Observational
Sponsor: Keiser University College of Chiropractic Medicine (Other)
Responsible Party: Principal Investigator, Maruti Gudavalli, Professor, Keiser University College of Chiropractic Medicine
Other Study IDs: IRB000OC18MG72
Record Dates: First submitted 2022-03-28; First posted 2022-06-02 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain; Cervical Pain; Neck Disorder; Low Back Disorder; Spine Injury
Keywords: back pain; neck pain; chiropractic; spine surgery; spine function
MeSH Terms: conditions — Low Back Pain; Neck Pain; Spinal Injuries; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cox chiropractic care — Manual distraction of spine in a prone position using specially assisted table
  Other Names: Flexion-distraction

SUMMARY:
Continued spinal pain following spine surgery is reported in up to 50% of patients. Disability and pain following spine surgery occurs. Repeat back surgery outcomes on Workers Compensation low back patients demonstrated larger number of patients did not come back to work. Such continued pain has biopsychosocial health relationships between the physical and the psychological and social factors that are associated with back pain and disability. Chiropractic consultation by post surgical continued pain (PSCP) patients occurs but the frequency, clinical treatment and outcomes of chiropractic treatment are not sufficiently documented. Conditions reported in continued pscp patients seeking care following spinal fusion are reported as sacroiliac joint pain, internal disc disruption, and zygapohyseal joint pain. Sacroiliac joint pain is more common after fusion, while internal disc disruption is more common in nonfusion patients. Very few studies are available on the outcomes of PSCP patients seen by chiropractic. This study proposes to investigate the clinical outcomes of PSCP patients presenting with pain in lumbar, thoracic, and cervical regions and had prior surgery in the respective regions, seeking care from field Doctors of Chiropractic (DCs) certified in Cox flexion distraction decompression procedures.

DETAILED DESCRIPTION:
Continued spinal pain following spine surgery is reported in up to 50% of patients. Disability and pain following spine surgery occurs. Repeat back surgery outcomes on Workers Compensation low back patients demonstrated larger number of patients did not come back to work. Such continued pain has biopsychosocial health relationships between the physical and the psychological and social factors that are associated with back pain and disability. Chiropractic consultation by post surgical continued pain (PSCP) patients occurs but the frequency, clinical treatment and outcomes of chiropractic treatment are not sufficiently documented. Conditions reported in continued pscp patients seeking care following spinal fusion are reported as sacroiliac joint pain, internal disc disruption, and zygapohyseal joint pain. Sacroiliac joint pain is more common after fusion, while internal disc disruption is more common in nonfusion patients. Very few studies are available on the outcomes of PSCP patients seen by chiropractic. This study proposes to investigate the clinical outcomes of PSCP patients presenting with pain in lumbar, thoracic, and cervical regions and had prior surgery in the respective regions, seeking care from field Doctors of Chiropractic (DCs) certified in Cox flexion distraction decompression procedures.

Research questions:

The specific aims of the study are:

Specific Aim 1: Descriptively document the subjective clinical outcomes (at visit one, at 3 months and at 12 months following intervention) regarding pain (using the VAS pain scale) and disability outcomes (using Roland Morris, Neck Disability Index, and PROMIS 29 questionnaires). Descriptively document the objective clinical outcome response (using a proforma exam form). This data will be collected regarding all patients who had undergone surgery to the lumbar, thoracic and/or cervical spines and choose to undergo care in the regions they had surgery with a Cox Certified Flexion-distraction decompression (FDD) practitioner. We expect to include 50 DCs and approximately 500 patients (an average of 10 patients per DC). Specific Aim 2: Descriptively document the treatment received during visits over a maximum of 3-month intervention. Determine the intervention details used by licensed Doctors of Chiropractic (DC) who are certified FDD and providing care to PSCP patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older.
* Have neck pain and associated radiating symptoms,thoracic pain, back pain and/or associated radiating symptoms and have undergone at least one spine surgery in the respective regions.
* Willing to undergo FDD chiropractic care in the painful regions of the spine.

Exclusion Criteria:

* Systemic arthropathies or other co-morbid conditions that may require care outside study and may affect ability to deliver study treatments or interfere with study ssessments;
* Inability to read or verbally comprehend English;
* Intention to move from the area during the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a prior surgery to the spine and reporting to chiropractic care for spinal pain
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
change in PROMISE 29 scores from initial visit to 3 months of treatment | baseline to 3 months
  Functional outcome of daily activities

SECONDARY OUTCOMES:
change in PROMISE 29 scores from initial visit to 12 months with 3 months of treatment | baseline to 12 months
  Functional outcome of daily activities
change in NDI scores from initial visit to 3 months of treatment | baseline to 3 months
  Functional outcome of daily activities
change in NDI scores from initial visit to 12 months with 3 months of treatment | baseline to 12 months
  Functional outcome of daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- Keiser University, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Any request for data will be shared according to University protocols